CLINICAL TRIAL: NCT05059353
Title: Open Label Clinical Trial to Study the Effectiveness and Safety of a Digitally Based Multidomain Intervention for Mild Cognitive Impairment
Brief Title: Effectiveness and Safety of a Digitally Based Multidomain Intervention for Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuroglee Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NG-001
Record Dates: First submitted 2021-08-30; First posted 2021-09-28 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This study comprises three study populations: patients with MCI, cognitively normal subjects, and caregivers of the patients with MCI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with MCI (Experimental)
  Interventions: Device: Digitally based multidomain intervention
- Cognitively Normal Subjects (Experimental)
  Interventions: Device: Digitally based multidomain intervention
- Caregivers of Patients with MCI (No Intervention)

INTERVENTIONS:
Device: Digitally based multidomain intervention — Education (5-10 mins). This session is to educate patients on instrumental activities of daily living such as the importance of companionship, medication, finance, home, travel, and kitchen safety. The content will be delivered using video and text-based material in English.
  Physical Activity (10 mins). This session includes activities such as brisk walking and yoga. Participants will be allowed to choose their preferred exercise option from the menu.
  Reminiscence Therapy (20 mins). This session includes recollection of events using directed questions, and a collection of photos from the past. Participants will be asked to share about any aspect related to the given topics using text or audio.
  Cognitive Games (20 mins). Participants will be asked to play games using their fingers to control characters on the screen to achieve goals. These games are designed to train different cognitive abilities, including attention, memory, executive functioning, and processing speed.
  Arms: Cognitively Normal Subjects; Patients with MCI

SUMMARY:
This study is designed to evaluate the preliminary effectiveness and safety of a digitally based multidomain intervention in patients with MCI. In addition, a portion of cognitively normal subjects and caregivers of patients with MCI will also be recruited as an exploratory cohort. We hope that the digital platform will improve the overall cognition and quality of life in patients with MCI.

DETAILED DESCRIPTION:
3 groups of participants will be recruited. For the participants in the MCI (group A) and cognitively normal subjects (group B), they will be provided with a digital tablet and a wearable device. The digital tablet will be pre-loaded with 10 modules, 1 module per week (1 hour) for 10 weeks to be completed at home. The wearable device will be used to track and collect physiological data.

For the caregivers of the patients with MCI (group C), they will be asked to complete a questionnaire during screening visit and follow-up visit, and to use the caregiver app during the intervention period.

ELIGIBILITY:
Patients with MCI Thirty (30) patients with MCI of the amnestic type (single or multi domain) will be recruited. MCI will be diagnosed using the Petersen's criteria and/or the NIA-AA criteria by cognitive neurologists.

Inclusion criteria:

1. Either male or female aged between 50 and 70 years (inclusive)
2. Diagnosis of amnestic MCI using the Petersen's criteria and/or the NIA-AA criteria
3. Clinical Dementia Rating (CDR) score of 0.5 and Mini-Mental State Examination (MMSE) >24
4. Education >6 years
5. Literate in English
6. Basic proficiency in using web-based applications/mobile platforms
7. Willing to give informed consent

Exclusion criteria:

1. Significant hearing or visual impairment
2. Significant systemic, neurological or psychiatric illness such as end stage renal failure, Parkinson's disease or major depression.
3. Participation in any pharmacological or non-pharmacological (interventional) clinical trial in the preceding 12 weeks

Cognitively Normal Subjects Ten (10) cognitively normal subjects will be recruited.

Inclusion criteria:

1. Either male or female aged between 50 and 70 years (inclusive)
2. CDR of 0 and MMSE > 27
3. Education >6 years
4. Literate in English
5. Basic proficiency in using web-based applications/mobile platforms
6. Willing to give informed consent

Exclusion criteria:

1. Significant hearing or visual impairment
2. Significant systemic, neurological or psychiatric illness such as end stage renal failure, Parkinson's disease or major depression.
3. Participation in any pharmacological or non-pharmacological clinical trial in the preceding 12 weeks

Caregivers of Patients with MCI Fifteen (15) caregivers of the 30 patients with MCI will be recruited.

Inclusion criteria:

1. Either male or female aged ≥21 years
2. Is the spouse or child of the patient and must spend at least 2 hours per week with the patient.
3. Must be healthy and not suffering from any serious systemic, neurological or psychiatric illness.
4. Literate in English
5. Willing to give informed consent Exclusion criteria: NA

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in processing speed | Baseline compared to Week 11
  Using Neuropsychological Test Battery (NTB) Processing Speed domain items (symbol digit modalities test, trail making test A, and Stroop test (condition 1 and 2) in patients with MCI
Change from baseline in executive functioning | Baseline compared to Week 11
  Using the NTB Executive Function domain items (digit span test, verbal fluency test, similarities test from Wechsler Adult Intelligence Scale IV (WAIS-IV) and trail making test B) in patients with MCI
Change from baseline in mood using the Depression Anxiety Stress Scales (DASS-21) in patients with MCI | Baseline compared to Week 11
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress.
  Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content.
  The scoring ranges from 0 to 3 per item. The higher the score, the greater the sense of depression, anxiety or stress.

SECONDARY OUTCOMES:
Change from baseline in overall cognition in patients with MCI | Baseline compared to Week 11
  Overall cognition is tested using the Neuropsychological Test Battery (NTB). Higher scores demonstrates better performance.
Change from baseline in QoL | Baseline compared to Week 11
  Using QOL-AD questionnaire in patients with MCI

CONTACTS AND LOCATIONS:
Overall Officials: Kok-Pin Ng, MBBS, Principal Investigator — National Neuroscience Institute
Locations (1):
- National Neuroscience Institute, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rykov YG, Ng KP, Patterson MD, Gangwar BA, Kandiah N. Predicting the severity of mood and neuropsychiatric symptoms from digital biomarkers using wearable physiological data and deep learning. Comput Biol Med. 2024 Sep;180:108959. doi: 10.1016/j.compbiomed.2024.108959. Epub 2024 Jul 31. PMID 39089109